CLINICAL TRIAL: NCT02839863
Title: Utrecht Cohort for Multiple Breast Cancer Intervention Studies and Long-term Evaluation - The UMBRELLA Cohort
Acronym: UMBRELLA
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Associate Professor, UMC Utrecht
Other Study IDs: NL52651.041.15
Record Dates: First submitted 2016-05-27; First posted 2016-07-21 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to better treatment options and earlier detection, survival rates of patients with breast cancer continue to increase. As such, (late) treatment toxicity, (long-term) quality of life and the cosmetic outcome are becoming more important. Also, many competing experimental interventions (e.g. treatment, lifestyle interventions) for breast cancer are being developed, all in need to be properly evaluated before being implemented in routine clinical care. Randomized Controlled Trials are the gold standard to do so, but they have shown many challenges, especially when applied in a cancer setting. The 'cohort multiple Randomized Controlled Trial (cmRCT)' design is a promising design for multiple (simultaneous) randomized evaluations of experimental interventions, with potential for increased recruitment, comparability and long-term outcomes as a standard.

By setting up UMBRELLA, as a prospective cohort according to the cmRCT design, the investigators aim to:

* provide an infrastructure for efficient, fast and pragmatic evaluation and implementation of experimental interventions
* gain insight into short and long-term treatment response, toxicity, complications, quality of life and survival of patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with breast cancer who undergo irradiation in the UMC Utrecht
* Informed consent - at least - for use of routinely collected clinical data and to fill out questionnaires.

Exclusion Criteria:

* Inability to understand the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients undergoing radiation treatment
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2053-10 (Estimated); Study Completion 2053-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Quality of Life at 10 years | 10 years
  Assesment of Health-related quality of life in breast cancer patients undergoing radiation

CONTACTS AND LOCATIONS:
Overall Officials: Helena M Verkooijen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Ziekenhuisgroep Twente, Almelo
  - Alrijne Ziekenhuis, Leiderdorp
  - St. Antonius Ziekenhuis, Nieuwegein
  - University Medical Center Utrecht, Utrecht